CLINICAL TRIAL: NCT04433598
Title: Effectiveness of Nutrition Education Intervention on Glycemic Control, and Other Diabetes-Related Outcomes of Patients With Type 2 Diabetes Mellitus In Basrah, Iraq.
Brief Title: Effectiveness of Nutrition Education Intervention on Glycemic Control (HbA1c)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Saman Agad Hashim, Nutritionist, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GS48062
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes; Diet, Healthy; Health Knowledge, Attitudes, Practice
Keywords: glycemic control; nutrition education; nutritional status; plate method; vegetables; health literacy; diabetes knowledge
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Intervention Model Description: This is a single-blinded parallel-randomized controlled trial (RCT) where type 2 diabetes mellitus (T2DM) participants were recruited in the study. The nutrition education intervention was consisted of four components: (1) the curriculum (twelve weekly sessions, 1 to 1.5 hrs. each); (2) follow-up sessions (bi-monthly, each lasting 1 to 1.5 hrs.); (3) Educational materials and (4) reminder calling before each session. The nutrition education intervention sessions will be presented in ten groups of ten participants (10 participants each day). The participants were backed up to bring a friend or a family member. The groups have been formed based on recruitment time; therefore, the nutrition education intervention sessions were staggered over the study period. This study has been presented the nutrition education intervention in the form of an easy and simple dietary plan management like plate method or consumption of vegetables before carbohydrates.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study was a single blinded parallel-randomized controlled trial, where the blinding assignment was after assignment of intervention. Participants, care providers and medical lab technicians (those assessing outcomes) at FDEMC were blinded after assignment to intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Education Intervention (Experimental): the participants the intervention group under went to Nutrition Education Intervention program were received the developed educational materials (pamphlets).
  Interventions: Behavioral: Nutrition Education Intervention
- Treatment as usual (No Intervention): the participants in the control group were received the usual medical care at their respective Center.The developed educational materials (pamphlets) were distributed at the end of the study.

INTERVENTIONS:
Behavioral: Nutrition Education Intervention — Each participant were interviewed by face- to- face using Arabic language, after 1 hour when they finish their assessment by medical doctors. The researcher was collected the data from the participants in a special room for 10-15 minutes, after only one hour of completing the necessary tests with the treating physician to allow participants to go for a meal before the nutrition education starts.12 classes (1:30 hour each session):- 100 participants / 5 days = 20 participants each class was offered twice per day to cover the number of participants and to enhance attendance for them can not attend at first morning. the classes was designed according to health belief model (HBM). The topics were about the type 2 diabetes and its complications,the benefits of diabetes plate and eating vegetables before carbohydrates.
  Arms: Nutrition Education Intervention

SUMMARY:
Aim: To evaluate the effect of nutrition education intervention (NEI) on glycemic control and other diabetes-related outcomes of patients with type 2 diabetes mellitus (T2DM), at a tertiary health Center, in Basrah, Iraq. Participants and setting: The study was involved 208 participants (20-64 years) diagnosed with T2DM at least 6 months before the study and had poorly controlled diabetes (HbA1c ≥ 7%). The study setting is the outpatient clinics at a tertiary health Center in Basrah, Iraq. Intervention: This randomized controlled trial design. The participants were allocated to either intervention group (IG), or control group (CG). A total sample size was 208 participants with T2DM (104 per group) to detect a 5% reduction in glycemic control (HbA1c), at visit time 1 (3 months after intervention) and visit time 2 (3 months after following up) and allowing 30% drop out rate. The intervention period is 22 weeks long with the following mechanisms: the curriculum (twelve weekly classes, 1 to 1.5 hrs. each); follow-up classes (one monthly each lasting 1 to 1.5 hrs.); nutrition education materials (pamphlets) and reminder calling before each session for IG. The participants in the CG received classes about diabetes and its complications with some advice related to physical activity on different days on IG. Besides, they received the same pamphlets at the end of the study. Both groups continued with the usual medical care at respective Center. The participants in the IG group received nutrition education classes. The classes are offered in the meeting hall in the center by face- to- face using the simple Arabic language, which utilized lecture method using PowerPoint presentations and whiteboard, lecture-discussion groups, and related videos. The nutrition education classes were administered by a nutritionist and a team of endocrinologists, and diabetes experts. The content and strategies utilized in the classes were based on Health Belief Model theory (HBM). Outcomes: the outcomes were evaluated at visit time 1 (at 12 weeks of intervention) and at visit time 2 (at 22 weeks of the follow-up period) for both groups. The outcomes were included HbA1c, metabolic parameters, nutritional status, HBM constructs, diabetes knowledge (DK), and health literacy (HL). It is assumed that the NEI will reduce the HbA1c levels by at least 0.5% at three months and the levels will be lower in IG compared with CG, and the lower levels will be continued at 22 weeks in IG.

DETAILED DESCRIPTION:
The aim of the study: To evaluate the effect of nutrition education intervention (NEI) on glycemic control and other diabetes-related outcomes of patients with type 2 diabetes mellitus (T2DM), at a tertiary health Center, in Basrah, Iraq. Specific objectives: (i) To describe and compare the glycemic control (HbA1c), socio-demographic status (age, gender, marital status, and employment), medical characteristics (duration of diabetes, family history, and blood pressure measures), nutritional status (anthropometric measurements, metabolic parameters, and dietary intake). Besides, lifestyle characteristics (physical activity level, smoking, and alcohol drinking), health belief model (HBM) constructs (susceptibility, severity, benefits, barriers, and self-efficacy), diabetes knowledge (DK), and health literacy (HL) level of patients with T2DM at baseline (T0), between intervention and control groups. (ii) To evaluate the effectiveness of NEI on glycemic control (HbA1c), medical characteristics, nutritional status, lifestyle characteristics, HBM constructs, DK, and HL level of patients within and between intervention and control groups at visit time 1 (T1), and visit time 2 (T2).

Participants and setting: The study was a parallel, randomized design, was conducted from June to December 2019, and involved 208 participants (20-64 years) diagnosed with T2DM at least 6 months before the study and had poorly controlled diabetes (HbA1c ≥ 7%). The study setting is the outpatient clinics at Faiha Specialized Diabetes, Endocrine, and Metabolism Centre (FDEMC), Basrah, Iraq. This study was involved in three phases based on the Generalized Model for Health Program Planning. Phase I included a cross-sectional study for need assessment among 280 participants with T2DM. The data that were collected included socio-demographic status, medical characteristics, nutritional status, lifestyle behavior, and health literacy. Phase II included the preparation and development of nutrition education materials based on HBM. Phase III was the randomized controlled trial among 208 participants with T2DM who attended the program were selected according to specific criteria. Participants aged between 20 and 64 years old, without hearing or vision problems and severe illnesses like cancers and renal failure were included in the study. The eligible participants signed the study consent form after the screening. The data were collected at baseline (T0), visit time 1 after 12 weeks of intervention (T1), and visit time 2 after 10 weeks of follow-up (T2). The institutional ethics committees approved the study and all participants provide their written consent before study enrollment.

Intervention: The participants were allocated using simple randomization to either intervention group (IG), or control group (CG). A total sample size was 208 participants with T2DM (104 per group) to detect a 5% reduction in glycemic control (HbA1c), at visit time 1 (3 months after intervention) and visit time 2 (3 months after following up) and allowing 30% drop out rate. The CONSORT report was followed up, wherever possible. The allocation was concealed using serially numbered opaque closed envelopes until intervention is assigned. The intervention period was 12 weeks long with the following mechanisms: the curriculum (twelve weekly classes, 1 to 1.5 hrs. each); follow-up classes (one monthly each lasting 1 to 1.5 hrs.); nutrition education materials (pamphlets) and reminder calling before each session for IG. The pamphlets were distributed for use at home as individual goal-setting activities. The participants were bucked up to bring a friend or a family member. While the follow-up period was 10 weeks long with the following mechanisms: monthly follow-up class, and reminder calling before each class for IG. The participants in the CG received classes about diabetes and its complications with some advice related to physical activity on different days on IG. Besides, they received the same educational materials (pamphlets) at the end of the study. Both groups continued with the usual medical care at respective Center. All the classes are offered in the meeting hall in the Center by face- to- face using the local Arabic language, which utilized the lecture method using PowerPoint presentations and whiteboard, lecture-discussion groups with household measurements to estimate the portion size and related videos or animations. The classes were concentrated on plate method and eating vegetables before carbohydrates as a simplified manner for participants with low HL. it were administered by a nutritionist and a team of endocrinologists, and diabetes experts. The content and strategies utilized in the intervention were based on Health Belief Model theory (HBM). Standardized questionnaires for data collection are considered as appropriate measures for the study outcomes and suitable for use it with the target patients.

Evaluation of intervention: The evaluations of the effectiveness of NEI were conducted at T1 and T2, on the following outcomes: (i) Clinical outcomes: HbA1c (%), lipid profile in mmol/L, and blood pressure in mmHg. (ii) Nutritional status: BMI in kg/m2, and dietary intake (energy intake in kilocalories per day, macronutrient intake in gram per day, vegetable and fruit intake in servings per day). (iii) Physical activity level in MET-min/week, and (iv) Potential behavior mediators: HBM constructs (susceptibility, severity, benefits, barriers, and self-efficacy), DK, and HL level. The outcome objective is to evaluate the changes between groups at T1 and T2 for HbA1c, lipid profile, and blood pressure, BMI, and dietary intake, physical activity level, HBM constructs, DK, and HL level. The study hypothesis: (i) intervention will reduce the HbA1c at T1 and these levels will be significantly lower in IG than CG, and these levels will remain significantly lower at T2. (ii) IG will have significantly better results in other diabetes-related outcomes that including nutritional status, physical activity level, blood pressure; HBM constructs, DK, and HL scores at T1, and these significantly improved results will maintain at T2 compared to CG. (iii) IG compared to CG will have significantly more patients who achieve a good HbA1c at T1 and will remain significantly lower at T2.

Data analysis: The general linear model (GLM) repeated measures ANCOVA was performed to measure the changes over time with the adjustment of significant differences at baseline as covariates. An intention-to-treat analysis (ITT) of all the outcomes of the study was achieved for non-adherence and missing outcomes. The level of significance was set at p < 0.05 for a two-tailed test.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a confirmed diagnosis of T2DM for at least one year prior to the study.
2. Iraqi participants aged 20-64 years.
3. Both males and females.
4. Current Basrah residents.
5. Arabic speaking participants due to the need for discussion in focus groups.
6. Participant are able to read or write.
7. Participants with marginal health literacy and above.

Exclusion Criteria:

1. Serious, severe illnesses (such as renal failure, myocardial infarction, cancer or surgery within the previous 4 weeks).
2. Intake of oral contraceptive drugs, steroid drugs or any hormones effects on blood glucose levels.
3. Participants with hearing or vision problems.
4. Heavy smokers (more than 40 cigarettes a day).
5. Pregnant women with gestational diabetes mellitus or lactating women.
6. Planning to move from the study area during the study period

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2019-06-09 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Glycemic control | From baseline to 12 weeks and 22 weeks
  Glycated Hemoglobin (HbA1c), taken from medical records (%) change

SECONDARY OUTCOMES:
Energy intake | From baseline to 12 weeks and 22 weeks
  Assessment of energy intake, using 3-days food record, mean energy intake (kcal/day)
Carbohydrates intake | From baseline to 12 weeks and 22 weeks
  Assessment of carbohydrates intake, using 3-days food record, mean carbohydrates intake (gram/day)
Protein intake | From baseline to 12 weeks and 22 weeks
  Assessment of protein intake, using 3-days food record, mean protein intake (gram/day)
Fat intake | From baseline to 12 weeks and 22 weeks
  Assessment of fat intake, using 3-days food record, mean fat intake (gram/day)
Dietary fiber intake | From baseline to 12 weeks and 22 weeks
  Assessment of dietary fiber intake, using 3-days food record, mean fiber intake (gram/day)
Fruit intake | From baseline to 12 weeks and 22 weeks
  Assessment of fruit intake, using 3-days food record, mean fruit intake (servings/day)
Vegetable intake | From baseline to 12 weeks and 22 weeks
  Assessment of vegetable intake, using 3-days food record, mean vegetable intake (servings/day)
Physical activity | From baseline to 12 weeks and 22 weeks
  Assessment of physical activity, using S-IPAQ questionnaire, mean physical activity (MET-min/week)
Waist circumference | From baseline to 12 weeks and 22 weeks
  Assessment of waist circumference, using tape measure, mean waist circumference (cm)
Weight | From baseline to 12 weeks and 22 weeks
  Assessment of weight, using weight scale, mean weight (kg)
BMI | From baseline to 12 weeks and 22 weeks
  Assessment of BMI, using weight and height scale to calculate BMI, mean BMI, (kg/m2)
Blood pressure | From baseline to 12 weeks and 22 weeks
  Assessment of systolic and diastolic blood pressure, taken from medical records, mean systolic and diastolic blood pressure (mmHg)
Fasting blood sugar | From baseline to 12 weeks and 22 weeks
  Assessment of fasting blood sugar, taken from medical records, mean fasting blood sugar (mmol/L)
Total cholesterol | From baseline to 12 weeks and 22 weeks
  Assessment of total cholesterol, taken from medical records, mean total cholesterol (mmol/L)
LDL-cholesterol | From baseline to 12 weeks and 22 weeks
  Assessment of LDL-cholesterol, taken from medical records, mean LDL-cholesterol (mmol/L)
HDL-cholesterol | From baseline to 12 weeks and 22 weeks
  Assessment of HDL-cholesterol, taken from medical records, mean HDL-cholesterol (mmol/L)
Triglycerides | From baseline to 12 weeks and 22 weeks
  Assessment of triglycerides, taken from medical records, mean triglycerides (mmol/L)
Health belief model (HBM) constructs | From baseline to 12 weeks and 22 weeks
  Assessment of HBM constructs, using questionnaire, mean HBM construct score (%)
Diabetes knowledge (DK) | From baseline to 12 weeks and 22 weeks
  Assessment of DK, using Michigan diabetes questionnaire (true and false version), mean DK score (%)
Health literacy (HL) | From baseline to 12 weeks and 22 weeks (%)
  Assessment of HL, using S-TOFHLA questionnaire, mean HL score

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Barakatun-Nisak M Yusof, PhD, Study Director — Universiti Putra Malaysia
Locations (1):
- Al-Faiha Diabetes Endocrine and Metabolism Center (FDEMC), Basra, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashim SA, Mohd Yusof BN, Abu Saad H, Ismail S, Hamdy O, Mansour AA. Effectiveness of simplified diabetes nutrition education on glycemic control and other diabetes-related outcomes in patients with type 2 diabetes mellitus. Clin Nutr ESPEN. 2021 Oct;45:141-149. doi: 10.1016/j.clnesp.2021.07.024. Epub 2021 Aug 3. PMID 34620310